CLINICAL TRIAL: NCT07015320
Title: The Behavioral and Alarm Therapy for Primary Monosymptomatic Nocturnal Enuresis , a Prospective Randomized Control Trial.
Brief Title: The Behavioral Therapy for Primary Monosymptomatic Nocturnal Enuresis
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelghany, lecturer, Cairo University
Other Study IDs: R408
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2023-01

CONDITIONS: Enuresis, Nocturnal
Keywords: nocturnal enuresis; behavioural therapy; urotherapy
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- urotherapy
  Interventions: Behavioral: urotherapy
- control
  Interventions: Behavioral: no intervention

INTERVENTIONS:
Behavioral: urotherapy — prompted and scheduled voiding, regular sleep timing, fluid and caffeine restriction and avoiding the cellular phones 2 hours before bedtime. If the child had constipation, it should be treated. In addition, alarm therapy was performed in the form of awaking the child every night by his parents after 1-2 hours from deep sleep to void then continue the sleep. The parents should be informed about the importance of their psychological support to their child by avoiding any punishment or embarrassment. Furthermore, the parents were asked to monitor their child's response by documenting the number of wet nights within the last month
  Groups: urotherapy
Behavioral: no intervention — no intervention
  Groups: control

SUMMARY:
A prospective randomized clinical study was conducted at Urology departments, faculties of medicine, Fayoum and Cairo Universities. All children either boys or girls between 4-4.5 years old presented with bedtime wetting despite good daytime urine control were included in the study. The children who were older than 4.5 years, had daytime voiding dysfunction, had !، behavioural disorders like attention deficient and hyperactivity disorder (ADHD) or other comorbidities like diabetes mellitus (DM) or congenital abnormalities were excluded from the study. In addition, those children whom parents refused to sign the consent of participation were also excluded. 120 children with primary monosymptomatic nocturnal enuresis (PMNE) were initially included in this study and randomized into two groups according to computer generated randomization. Group A (early therapy) included initially 60 child who had done behavioural and alarm therapy from the start of the study regularly till the age of 5.5 years and Group B (deferred therapy) included 60 child who waited without therapy till age of 5 years, then they started the behavioural and alarm therapy regularly for 6 months. They were interviewed at urology clinics in Fayoum and Cairo Universities in Egypt. The behavioural therapy was in the form of prompted and scheduled voiding, regular sleep timing, fluid and caffeine restriction and avoiding the cellular phones 2 hours before bedtime. If the child had constipation, it should be treated. In addition, alarm therapy was performed in the form of awaking the child every night by his parents after 1-2 hours from deep sleep to void then continue the sleep. The parents should be informed about the importance of their psychological support I to their child by avoiding any punishment or embarrassment. Furthermore, the parents were asked to monitor their child's response by documenting the number of wet nights within the last 4 month. All children were then evaluated at the age of 5 and 5.5 years using the following outcomes through the last month before the visit: complete response (0 wet nights), > 80 % stoppage of bedwetting (< 6 wet nights), 50-80 % stoppage of bedwetting (6-15 wet nights) and < 50 % stoppage of bedwetting (> 15 wet nights).

DETAILED DESCRIPTION:
A prospective randomized clinical study was conducted at Urology departments, faculties of medicine, Fayoum and Cairo Universities. All children either boys or girls between 4-4.5 years old presented with bedtime wetting despite good daytime urine control were included in the study. The children who were older than 4.5 years, had daytime voiding dysfunction, had behavioural disorders like attention deficient and hyperactivity disorder (ADHD) or other comorbidities like diabetes mellitus (DM) or congenital abnormalities were excluded from the study. In addition, those children whom parents refused to sign the consent of participation were also excluded. 120 children with primary monosymptomatic nocturnal enuresis (PMNE) were initially included in this study. They were randomized into two groups according to computer generated randomization. Group A (early therapy) included initially 60 child who had done behavioural and alarm therapy from the start of the study regularly till the age of 5.5 years and Group B (deferred therapy) included 60 child who waited without therapy till age of 5 years, then they started the behavioural and alarm therapy regularly for 6 months. They were interviewed at urology clinics in Fayoum and Cairo Universities in Egypt. The behavioural therapy was in the form of prompted and scheduled voiding, regular sleep timing, fluid and caffeine restriction and avoiding the cellular phones 2 hours before bedtime. If the child had constipation, it should be treated. In addition, alarm therapy was performed in the form of awaking the child every night by his parents after 1-2 hours from deep sleep to void then continue the sleep. The parents should be informed about the importance of their psychological support to their child by avoiding any punishment or embarrassment. Furthermore, the parents were asked to monitor their child's response by documenting the number of wet nights within the last 4 month. All children were then evaluated at the age of 5 and 5.5 years using the following outcomes through the last month before the visit: complete response (0 wet nights), > 80 % stoppage of bedwetting (< 6 wet nights), 50-80 % stoppage of bedwetting (6-15 wet nights) and < 50 % stoppage of bedwetting (> 15 wet nights).

ELIGIBILITY:
Inclusion Criteria:

* PMNE

Exclusion Criteria:

* neurogenic bladder

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: PMNE
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
bed wetting | 6 months
  complete response (0 wet nights), > 80 % stoppage of bedwetting (< 6 wet nights), 50-80 % stoppage of bedwetting (6-15 wet nights) and < 50 % stoppage of bedwetting (> 15 wet nights).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt